CLINICAL TRIAL: NCT03899415
Title: TCR-Redirected T Cells Therapy in Patient With HBV Related HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Lion TCR Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-3-1
Record Dates: First submitted 2019-01-17; First posted 2019-04-02 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-Redirected T Cells (Experimental): HBV antigen specific TCR redirected T cells
  Interventions: Biological: TCR redirected T cells

INTERVENTIONS:
Biological: TCR redirected T cells — HBV antigen specific TCR redirected T cell Infusions. Subjects will receive 1x10^4 - 5x10^6 TCR redirected T cells by IV infusion.

SUMMARY:
This is a single center. single arm, open-label study to determine the safety and clinical benefit of TCR-redirected T cell therapy in patient with HBV related HCC post hepatectomy or radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Expression of the specific human leukocyte antigen (HLA) class I profile
2. Hepatocellular carcinoma (HCC) with positive test for hepatitis B virus surface antigen (HBsAg)
3. BCLC stage C
4. At least 1 month after surgical intervention or 2 weeks after TACE (may include other type of resection/ablation) No major post-operative complication
5. Laboratory criteria:

   1. Liver function: Child A, ALT < 200 U/L, AST < 200 U/L, Tbil < 17.1umol/L
   2. Renal Function: Creatinine clearance ≥ 60ml/minute
   3. Cardiac Function: No abnormality in cardiac enzyme and ECG
   4. Pulmonary Function (Lung): No abnormality in chest X-ray
6. Sexually active subjects must be willing to use an acceptable method of contraception
7. Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures

Exclusion Criteria:

1. Subject experiencing acute infection or gastric bleeding within 30 days
2. Mid to late stage cirrhosis, i.e. Child-Pugh Score ≥ 7
3. Known history of testing positive for human immunodeficiency virus (HIV)
4. Other liver complications, including alcoholic liver disease, non-alcoholic autoimmune liver disease, drug induced liver disease
5. Serious systemic conditions, such as mental illness, cerebrovascular disease, coronary heart disease, diabetes, epilepsy
6. Women who are pregnant or breast-feeding
7. History of allergic reaction to blood products or investigational products
8. History of chronic alcoholism or drug abuse/addiction
9. Require systemic medications, such as steroids during the period of study drug administration
10. Exposure to any cell therapy such as, but not limited to NK, CIK, DC, CTL, stem cells therapy 6 months prior to study drug administration
11. Use of any investigational product (IP) or investigational medical device
12. Any condition which could jeopardize the safety of the patient and his/her compliance in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-20 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation based in Incidences of adverse events/serious adverse events | Up to 1 month after the last infusion
  Review the safety profile of T-Cell Therapy by assessing adverse/serious adverse events reported.

SECONDARY OUTCOMES:
Overall Response Rate | Start of Treatment until first documented CR or PR, assessed up to 56 treatment weeks (protocol-defined treatment duration is until disease progression, death, or loss to follow up, whichever came first)
  Tumour assessment will be according to mRECIST v1.1. This is based on percentage of participants with Complete Response (CR) and Partial Response (PR) according to mRECIST v1.1 from baseline.
Overall survival rate | Up to 5 years from the last infusion
  Overall Survival (OS) defined as the time from randomisation until death by any cause. Participants will be followed up for survival follow up for at least five years.

CONTACTS AND LOCATIONS:
Overall Officials: Fusheng Wang, MD, Principal Investigator — Beijing 302 Hospital of China
Locations (1):
- Beijing 302 Hospital of China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meng F, Zhao J, Tan AT, Hu W, Wang SY, Jin J, Wu J, Li Y, Shi L, Fu JL, Yu S, Shen Y, Liu L, Luan J, Shi M, Xie Y, Zhou CB, Wong RW, Lu-En W, Koh S, Bertoletti A, Wang T, Zhang JY, Wang FS. Immunotherapy of HBV-related advanced hepatocellular carcinoma with short-term HBV-specific TCR expressed T cells: results of dose escalation, phase I trial. Hepatol Int. 2021 Dec;15(6):1402-1412. doi: 10.1007/s12072-021-10250-2. Epub 2021 Nov 30. PMID 34850325